CLINICAL TRIAL: NCT06115174
Title: Clinical Study Evaluating the Anticancer Effect of Pentoxiphylline in Patients With Metastatic Colorectal Cancer
Acronym: CRC - PTX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nada Abu Eleneen Darwiesh Ibrahim, Bachelor of Clinical Pharmacy (2021) - Faculty of Pharmacy - Mansoura University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pentoxiphylline in CRC
Record Dates: First submitted 2023-10-13; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Pentoxifylline; Folfox protocol; XELOX; Antibodies, Monoclonal

STUDY DESIGN:
Intervention Model Description: The design of this study is a randomized, controlled parallel clinical trial which will be conducted on 44 patients with metastatic colorectal cancer. The duration of the study will be one year to determine progression free survival (PFS) and the overall survival (OS). Patients will be recruited from Medical Oncology Department, Oncology Centre, Mansoura University, Mansoura, Egypt. The patients will be randomized using sealed envelope method into the following two groups:
  Group I (Control group; n=22) which will receive FOLFOX (leucovorin, fluorouracil, oxaliplatin) or XELOX (oxaliplatin + capecitabine) ± target therapy (Bevacizumab).
  Group II: (Pentoxiphylline group; n=22) which will receive the same FOLFOX or XELOX regimen ± target therapy (Bevacizumab) in addition to Pentoxiphylline 400 mg twice daily.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People not recieving the drug (Other): (Control group; n=22) which will receive FOLFOX (leucovorin, fluorouracil, oxaliplatin) or XELOX (oxaliplatin + capecitabine) ± target therapy (Bevacizumab).
  Interventions: Radiation: FOLFOX; Radiation: XELOX; Drug: Monoclonal antibodies (target therapy)
- People recieving the drug (Active Comparator): (Pentoxiphylline group; n=22) which will receive the same FOLFOX (leucovorin, fluorouracil, oxaliplatin) or XELOX regimen (oxaliplatin + capecitabine) ± target therapy (Bevacizumab) in addition to Pentoxiphylline 400 mg twice daily.
  Interventions: Drug: Pentoxifylline; Radiation: FOLFOX; Radiation: XELOX; Drug: Monoclonal antibodies (target therapy)

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline (PTX) is a methylxanthine derivative that is commercially available in the name of Trental. It is currently used for management of peripheral vascular diseases. Its postulated mechanism of action is thought to be mediated through reducing blood viscosity and enhancing RBCs flexibility. However, it has been shown that PTX also may potentially be used in the anticancer therapy [15].
  The studies demonstrated the potential effects of pentoxifylline on angiogenesis inhibition. It can affect the release and function of some predominantly proangiogenic vascular endothelial growth factors. Specifically, the release of the VEGF family of pro-angiogenesis factors (notably VEGF-A and VEGF-C) [16]. Furthermore, the mechanism by which pentoxifylline inhibits angiogenesis may be through the inhibition of activation of STAT3 which contributes to tumor cell survival by regulating the expression of metastatic genes, MMPs, serine protease uPA and potent angiogenic genes [17].
  Arms: People recieving the drug
Radiation: FOLFOX — (leucovorin, fluorouracil, oxaliplatin)
Radiation: XELOX — (oxaliplatin + capecitabine)
Drug: Monoclonal antibodies (target therapy) — target therapy (Bevacizumab).

SUMMARY:
The aim of this work is to assess the antitumor effect of Pentoxiphylline in patients with metastatic colorectal cancer receiving stomatal chemotherapy ± targeted therapy.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) ranks as the third most common cancer globally and second in terms of mortality. Although CRC incidence rates are higher in high-income compared with low-to-middle-income countries (LMICs), mortality is higher in LMICs. And although more than 90% of CRC cases are diagnosed in individuals over age 55, CRC incidence is rising in younger populations. For example, Egypt, Saudi Arabia, the Philippines, and Iran have CRC incidence rates in individuals under age 40 of 38%, 21%, 17%, and 15%-35%, respectively. This is compared with only 2%-8% of new cases in the U.S. and the European Union in individuals in this age bracket. Along with the high incidence rate of CRC in individuals under age 40 in Egypt, CRC is diagnosed at more advanced stages in these younger Egyptians. CRC survival is highly dependent upon the stage of disease at diagnosis and typically ranges from a 90% 5-year survival rate for cancers detected at the localized stage to 14% for individuals diagnosed with distant metastatic cancer.

Apoptosis may occur via two major interconnected pathways: the extrinsic or death receptor-mediated pathway, which is activated by the binding of specific ligands (such as FasL, TNF-α and TRAIL) to the receptors of cell surfaces; and the intrinsic or mitochondrial-mediated pathway, which is regulated through proteins of the Bcl-2 family and triggered either by the loss of growth factor signals or in response to genotoxic stress. Therefore the replication of cells with DNA damage is generally avoided because harmful genomic alterations typically induce the activation of apoptosis. It has been widely accepted that alterations in the physiologic response to DNA damage can facilitate the accumulation of oncogenic mutations; this accumulation may eventually lead to the development of neoplasia.

Angiogenesis is a complex process by which new blood vessels are formed from endothelial precursor. It is a critical step in cancer progression and is considered one of the hallmarks of cancer. This process is mediated through a group of ligands and receptors that work in tight regulation. A group of glycoproteins, including the VEGFs (VEGF-A, VEGF-B, VEGF-C, and VEGF-D) and the placental growth factor (PIGF), act as effectors of angiogenesis. These factors interact with three VEGF receptors (VEGFR- 1, VEGFR-2, and VEGFR-3) and two neuropilin co-receptors (NRP1 and NRP2). The VEGF-A gene consists of eight exons with splice variants forming different isoforms, namely, VEGFA121, VEGFA165, VEGFA189, and VEGFA209; VEGFA165 is the most biologically active of these isoforms [14]. The VEGFRs are tyrosine kinase receptors that are primarily located in the vascular endothelial cells. The binding of VEGF-A to VEGFR-2 is believed to be the most important activator of angiogenesis.

Pentoxifylline (PTX) is a methylxanthine derivative that is commercially available in the name of Trental. It is currently used for management of peripheral vascular diseases. Its postulated mechanism of action is thought to be mediated through reducing blood viscosity and enhancing RBCs flexibility. However, it has been shown that PTX also may potentially be used in the anticancer therapy.

The studies demonstrated the potential effects of pentoxifylline on angiogenesis inhibition. It can affect the release and function of some predominantly proangiogenic vascular endothelial growth factors. Specifically, the release of the VEGF family of pro-angiogenesis factors (notably VEGF-A and VEGF-C) [16]. Furthermore, the mechanism by which pentoxifylline inhibits angiogenesis may be through the inhibition of activation of STAT3 which contributes to tumor cell survival by regulating the expression of metastatic genes, MMPs, serine protease uPA and potent angiogenic genes.

In addition, PTX has also the ability to induce apoptosis and potentiate the apoptotic effects of chemotherapy in several cancer types, one major mechanism is through activation of the caspase-dependent apoptosis that is accompanied by a decrease in kappa B-alpha- phosphorylation and up-regulation of the pro-apoptotic genes Bax, Bad, Bak, and caspases- 3,

-8, and -9.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically and/or radiologically confirmed diagnosis of metastatic colorectal carcinoma.
* Both genders.
* Age ≥ 18 years old, and ≤ 75 years old.
* Performance status 0-1 according to the Eastern Cooperative Oncology Group (ECOG).
* Patients with adequate hematologic parameters (white blood cell count

  ≥3000/mm3, granulocytes ≥1500/mm3, platelets ≥100,000/mm3, hemoglobin ≥ 8 gm/l).
* Patients with adequate renal functions (serum creatinine ≤1.5 mg/dL).
* Patients with adequate hepatic functions (bilirubin ≤1.5 mg/dL or albumin ≥3 g/dL).

Exclusion Criteria:

* Patients with active liver diseases (chronic viral hepatitis, autoimmune hepatitis, alcoholic hepatitis, Wilson's disease, hemochromatosis, or cirrhosis).
* Patients with brain metastasis.
* Patients with active infection.
* Patients on chronic use of corticosteroids.
* Patients receiving blood thinning agents(aspirin, clopidogrel, warfarin)
* Patients with other malignancy (synchronous, or metachronous)
* Prior exposure to neurotoxic drugs (oxaliplatin, cisplatin, vincristine, paclitaxel, or docetaxel, INH) for at least 6 months prior the study treatment.
* Evidence of pre-existing peripheral neuropathy resulting from another reason (diabetes, brain tumor, brain trauma, HCV, thyroid disorder).
* Patients with diabetes and other conditions that predispose to neuropathy as hypothyroidism, autoimmune diseases, hepatitis C.
* History of known allergy to oxaliplatin or other platinum agents.
* Patients with moderate and severe renal impairment (CrCl <50 ml/min) or serum creatinine >1.5 mg/dl.
* Pregnant and breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of RECIST between the two groups. | one year
  Difference in response rate (RECIST) between the control and drug groups.
Change in the serum concentration of the measured biological markers. | one year
Difference in progression free survival 'PFS' between the two groups | One year.
Difference in overall survival 'OS' between the two groups. | One year.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Mohammed, Professor, Study Chair — Tanta University; Dalia Refaat, Assistant Professor, Study Chair — Tanta University; Sherif Refaat, Lecturer, Study Chair — Oncology Centre - Faculty of Medicine - Mansoura University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Ferlay J, Colombet M, Soerjomataram I, Dyba T, Randi G, Bettio M, Gavin A, Visser O, Bray F. Cancer incidence and mortality patterns in Europe: Estimates for 40 countries and 25 major cancers in 2018. Eur J Cancer. 2018 Nov;103:356-387. doi: 10.1016/j.ejca.2018.07.005. Epub 2018 Aug 9. PMID 30100160
- [Background] Arnold M, Sierra MS, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global patterns and trends in colorectal cancer incidence and mortality. Gut. 2017 Apr;66(4):683-691. doi: 10.1136/gutjnl-2015-310912. Epub 2016 Jan 27. PMID 26818619
- [Background] Schreuders EH, Ruco A, Rabeneck L, Schoen RE, Sung JJ, Young GP, Kuipers EJ. Colorectal cancer screening: a global overview of existing programmes. Gut. 2015 Oct;64(10):1637-49. doi: 10.1136/gutjnl-2014-309086. Epub 2015 Jun 3. PMID 26041752
- [Background] Sankaranarayanan R. Screening for cancer in low- and middle-income countries. Ann Glob Health. 2014 Sep-Oct;80(5):412-7. doi: 10.1016/j.aogh.2014.09.014. PMID 25512156
- [Background] Haggar FA, Boushey RP. Colorectal cancer epidemiology: incidence, mortality, survival, and risk factors. Clin Colon Rectal Surg. 2009 Nov;22(4):191-7. doi: 10.1055/s-0029-1242458. PMID 21037809
- [Background] Marley AR, Nan H. Epidemiology of colorectal cancer. Int J Mol Epidemiol Genet. 2016 Sep 30;7(3):105-114. eCollection 2016. PMID 27766137
- [Background] Vuik FE, Nieuwenburg SA, Bardou M, Lansdorp-Vogelaar I, Dinis-Ribeiro M, Bento MJ, Zadnik V, Pellise M, Esteban L, Kaminski MF, Suchanek S, Ngo O, Majek O, Leja M, Kuipers EJ, Spaander MC. Increasing incidence of colorectal cancer in young adults in Europe over the last 25 years. Gut. 2019 Oct;68(10):1820-1826. doi: 10.1136/gutjnl-2018-317592. Epub 2019 May 16. PMID 31097539
- [Background] Abou-Zeid AA, Khafagy W, Marzouk DM, Alaa A, Mostafa I, Ela MA. Colorectal cancer in Egypt. Dis Colon Rectum. 2002 Sep;45(9):1255-60. doi: 10.1007/s10350-004-6401-z. PMID 12352245
- [Background] Gado A, Ebeid B, Abdelmohsen A, et al. Colorectal cancer in Egypt is commoner in young people: Is this cause for alarm? Alexandria J Med. 2014; 50:197-201.
- [Background] Metwally IH, Shetiwy M, Elalfy AF, et al. Epidemiology and survival of colon cancer among Egyptians: A retrospective study. J Coloproctol. 2018;38:24-29.
- [Background] American Cancer Society: Treatment of Colon Cancer, by Stage. 2020. Available at https://www.cancer.org/cancer/colon-rectal-cancer/ treating/by-stage- colon.html.
- [Background] Alcaide J, Funez R, Rueda A, Perez-Ruiz E, Pereda T, Rodrigo I, Covenas R, Munoz M, Redondo M. The role and prognostic value of apoptosis in colorectal carcinoma. BMC Clin Pathol. 2013 Oct 10;13(1):24. doi: 10.1186/1472-6890-13-24. PMID 24106912
- [Background] Mousa L, Salem ME, Mikhail S. Biomarkers of Angiogenesis in Colorectal Cancer. Biomark Cancer. 2015 Oct 27;7(Suppl 1):13-9. doi: 10.4137/BIC.S25250. eCollection 2015. PMID 26543385
- [Background] Meirovitz A, Baider L, Peretz T, Stephanos S, Barak V. Effect of pentoxifylline on colon cancer patients treated with chemotherapy (Part I). Tumour Biol. 2021;43(1):341-349. doi: 10.3233/TUB-211533. PMID 34957976
- [Background] Khoury W, Trus R, Chen X, Baghaie L, Clark M, Szewczuk MR, El-Diasty M. Parsimonious Effect of Pentoxifylline on Angiogenesis: A Novel Pentoxifylline-Biased Adenosine G Protein-Coupled Receptor Signaling Platform. Cells. 2023 Apr 20;12(8):1199. doi: 10.3390/cells12081199. PMID 37190108
- [Background] Dhumale P, Nikam Y, Gude R. Pentoxifylline: A potent inhibitor of angiogenesis via blocking STAT3 signaling in B16F10 melanoma. Int J Tumor Ther. 2013 ;2:1-9.
- [Background] Al-Husein BA, Mhaidat NM, Alzoubi KH, et al. Pentoxifylline induces caspase- dependent apoptosis in colorectal cancer cells. Inform Med Unlocked. 2022;31:100997
- [Background] Cuituny-Romero AK1, Onofre-Castillo J. Radiological evaluation, with RECIST criteria of treatment response of non-microcytic lung cancer. Anales de Radiologia México. 2015;14:31-42.